CLINICAL TRIAL: NCT00201383
Title: Phase III Study Of Post-Operative Adjuvant Concurrent Chemoradiotherapy For High Risk Oral Cavity Squamous Cell Carcinoma Patients
Brief Title: Post-Operative Adjuvant Concurrent Chemoradiotherapy For High Risk Oral Cavity Squamous Cell Carcinoma Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Changhua Christian Hospital (Other); China Medical University Hospital (Other); Buddhist Tzu Chi General Hospital (Other); Mackay Memorial Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other); Chi Mei Medical Hospital (Other); Kaohsiung Veterans General Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2399
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-01

CONDITIONS: Oral Cavity; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — Cisplatin

INTERVENTIONS:
Drug: cisplatin

SUMMARY:
The purpose of this study is to confirm the value of concurrent chemoradiotherapy in improving the locoregional control and survival of patients with resected locally advanced HNSCC, a phase III randomized study is proposed. The population studied in this trial is limited to patients of oral cavity cancer; this could reduce the confounding factor of varying prognosis in patients of different primary sites of HNSCC.

DETAILED DESCRIPTION:
Potentially resectable Stage III or IV squamous cell carcinomas of the head and neck (HNSCC) are treated by operation and adjuvant radiotherapy. The 5-year survival rate is approximating 30%. Recurrence typically occurs within 3 years, 60-80% in locoregional sites, and 20-30% systemically. Patients who are found to have tumors at the margins of surgical specimens far particularly poorly.

Chemotherapy has been added in the hope to improve this situation. Induction and adjuvant chemotherapy has resulted in a decrease in the appearance of systemic metastases in most trials, but has not improved locoregional control and survival.

For cases with unresectable head and neck cancers, concurrent chemoradiotherapy appears to have improved locoregional control, disease-free survival, and possibly overall survival, as compared to radiotherapy alone. Bachaud et al. reported a randomized trial of postoperative cisplatin and radiotherapy vs. radiotherapy alone for patients with Stage III or IV head and neck cancer. Cisplatin was administered 50 mg weekly during radiotherapy. There was a significant improvement in locoregional control (70% vs. 55%) as well as overall survival (median 36m vs. 20m) in patients who received concurrent chemoradiotherapy. Al-Sarraf et al. also reported a phase II concurrent chemoradiotherapy trial, using cisplatin 100 mg/m2 every three weeks. Based on comparison with similar patients treated in a prior RTOG trial, they conclude that postoperative radiotherapy with concurrent cisplatin may improve locoregional control rates10. The superiority of adjuvant concurrent chemoradiotherapy (CCRT) to RT alone or sequential adjuvant RT and chemotherapy has been further confirmed in an analysis of data of RTOG 85-03 and RTOG 88-24. Comparing high-risk patients of RTOG 85-03 with prognostically similar patients from RTOG 88-24, the data suggest that sequential surgery, RT, and chemotherapy produced better locoregional control than surgery plus RT, but that surgery followed by CCRT produced even higher locoregional control. Independent of the differences in the amount of RT delivered, the Cox proportional hazards model suggests that the addition of CCRT resulted in a 50% decrease in locoregional relapse rates compared with surgery plus postoperative RT with no chemotherapy. The reduction in mortality was 18%.

Although CCRT may be better than RT alone or sequential treatment, the 3 year survival in both adjuvant CCRT studies were only around 50%. Is more aggressive treatment warranted? Tolerance to CCRT is a major concern. In the French study, severe acute toxicity occurred in 18% of RT only patients and 41% of patients received CCRT. In the RTOG 88-24 trial, severe and life-threatening toxicities occurred in 20% and 12% of patients, respectively; the most common drug-related toxicities were leukopenia, anemia, nausea, and vomiting . Theoretically, to optimize CCRT, continuous presence of chemotherapeutic drug or drug effect is necessary to maximize the effect of radiosensitization. For radiosensitization purpose, daily chemotherapy may be better than weekly and weekly may be better than tri-weekly. French study used weekly cisplatin with a dose of 30 mg/m2. RTOG 88-24 used different treatment dose and schedule 100 mg/m2 of cisplatin on radiotherapy days 1, 23 and 43. We choose weekly for convenience and hope this can increase the recruitment of patients. In the pilot study, we observed a remarkable toxicity with this treatment schedule. Considering the remarkable toxicity reported and our preliminary experience, more drugs, higher dosage, or extended schedule may not be justified.

ELIGIBILITY:
Inclusion Criteria:

Clinically free of disease after having undergone surgery for histologically confirmed primary keratinizing SCC of the oral cavity.

buccal mucosa upper lip (140.3) lower lip (140.4) cheek (145.0) retromolar area (145.6) bucco-alveolar sulci upper and lower (145.1) oral tongue dorsum (141.1) lateral border (141.2) inferior surface (141.3)

With any one of the risk factors of recurrence listed below:

Nodal extracapsular spread of disease (ECS) Number of positive node > 2 Perineural involvement Lymphovascular emboli/permeation in resected surgical specimen Histologically positive surgical margin

Exclusion Criteria:

Karnofsky performance status of <50 Concurrent or previous second primary cancer (excluding non-melanoma skin cancer) Gross residual disease following surgery Distant metastasis before or at the time of adjuvant treatment Serum creatinine > 1.4 mg/dl, WBC <3500/mm3, platelet <100,000/mm3

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161
Dates: Start 1999-10; Study Completion 2009-08

PRIMARY OUTCOMES:
RT versus RT plus CT in effect on local control and survival of patients of oral cavity cancer after curative operation.

SECONDARY OUTCOMES:
the acute and chronic toxicity of RT versus RT plus CT in patients of oral cavity cancer after curative operation.

CONTACTS AND LOCATIONS:
Overall Officials: Mow-Ming Hsu, MD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- See also: Related Info — http://www.nhri.org.tw